CLINICAL TRIAL: NCT04819139
Title: Interaction Between Position Sense, Force Control and Pain Intensity in Basal Thumb Osteoarthritis. A Cross-sectional Study.
Brief Title: Position Sense, Force Control and Pain Intensity in Basal Thumb Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Raquel Cantero-Téllez, Principal investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-THUMB-1
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Thumb Osteoarthritis; Proprioceptive Disorders; Pain, Chronic
MeSH Terms: conditions — Somatosensory Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thumb exercises +orthosis (Active Comparator): Participants will be instructed to perform daily exercises grouped in 3 sets of 10 repetitions in the absence of pain for 4 weeks. If the patient experienced pain, the number of repetitions dropped sequentially until the exercise was performed pain free. Exercises consisted of active - resistive exercises for the first dorsal interosseous (FDI) muscle, manual distraction of the CMC joint and relaxation of the adductor thumb muscle. Each participant will also engaged in a one month re-education/joint protection program for thumb use during ADL's and completed a weekly record sheet for monitoring purposes.
  In addiction, they will received a "thumb whale" orthosis to wear at night and during ADL's as needed for pain.
  Interventions: Other: Active Excersises; Other: Reeducation ADL; Other: Joint protection
- Thumb exercises +orthosis+ proprioceptive program exercises (Experimental): Participants will be instructed to perform daily exercises grouped in 3 sets of 10 repetitions in the absence of pain for 4 weeks. If the patient experienced pain, the number of repetitions dropped sequentially until the exercise was performed pain free. Exercises consisted of active - resistive exercises for the first dorsal interosseous (FDI) muscle, manual distraction of the CMC joint and relaxation of the adductor thumb muscle. Each participant will also engaged in a one month re-education/joint protection program for thumb use during ADL's and completed a weekly record sheet for monitoring purposes.
  In addiction, they will received a "thumb whale" orthosis to wear at night and during ADL's as needed for pain. In addiction, patients will received a proprioceptive program exercises using also a online program with a laptop.
  Interventions: Other: Active Excersises; Other: Reeducation ADL; Other: Joint protection; Other: Proprioception exercises

INTERVENTIONS:
Other: Active Excersises — Active thumb exercises
Other: Reeducation ADL — Reeducation in the activities daily life
Other: Joint protection — Used of a thumb orthosis
Other: Proprioception exercises — Specific proprioception exercises
  Arms: Thumb exercises +orthosis+ proprioceptive program exercises

SUMMARY:
In practice, a single test is used to quantify thumb proprioception. Previous studies have found a decrease in joint position sense (JPS) and force sense (FS) in patients diagnosis of thumb carpometacarpal osteoarthritis, but no correlation have been stabilize between JPS, FS and pain intensity perceived by the patient during activity daily life (ADL).

The goal of the study is compared joint position error (JPE) with joint force sense error (JFSE) in subjects with carpometacarpal (CMC) joint osteoarthritis and investigated a possible correlation between thumb pain intensity and thumb proprioception in patients with CMC joint OA.

DETAILED DESCRIPTION:
Forty-five subjects over 18 with thumb CMC joint OA in the dominant hand grade 1-3 according o the Eaton Classification Stage will be evaluated for thumb active joint position sense (JPS) test and Force sense test to measure proprioception function. For measurement of JPS, the subjects will blindfolded and repositioned their thumb to a target position, which will be determined by the examiner previously. For force sense, participants will should reproduce pinch force measure with dynamometer. The severity of pain with activity will be measured according to the visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years; Diagnosis of grade I, II or II thumb CMC joint OA in their dominant hand according to the Eaton Classification Stage; A minimum pain rating of 4/10 on the Visual Analogue Scale (VAS) during activities of daily living (ADLs) at the time of the initial evaluation; Ability to read and understand the patient information sheets and exercises

Exclusion Criteria:

* Neurological disorder affecting the upper limb; Treatment for hand or thumb pain in the same limb in the last 6 months (including injections to the wrist, fingers, or thumb); Fracture or significant hand injury; Previous surgery to the wrist or hand; Hand/finger tenosynovitis; Dupuytren disease; Cognitive impairment that inhibited an understanding of the informed consent and exercise program; Fixed thumb adduction contracture or blindness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | baseline - 2 days
  Pain intensity will be measured according to the visual analog scale (VAS). The VAS scale is a unidimensional measure of pain intensity and is widely used in adult populations, including those with rheumatic diseases. Sensitivity and reliability of the instrument are well defined including sensitivity to change in pain for patients with chronic inflammatory or degenerative joint pain

SECONDARY OUTCOMES:
JPS | baseline - 2 days
  For measurement of JPS, the subjects were blindfolded and repositioned their thumb to a target position, which was determined by the examiner previously
FS | baseline- 2 days
  For force sense, participants should reproduce pinch force measure with dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Cantero-Téllez, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No